CLINICAL TRIAL: NCT06736015
Title: Use of Myo-inositol and Selenium in Patients with Indeterminate Thyroid Nodules (TIR3A)
Brief Title: Myo-inositol and Selenium in Indeterminate Thyroid Nodules (TIR3a)
Acronym: MYOSEL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Principal Investigator, Marialuisa Appetecchia, Chief of the Oncological Endocrinology Unit, Regina Elena Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RS39/IRE/23(2869)
Record Dates: First submitted 2024-12-05; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Thyroid Nodule
Keywords: TIR3A; indeterminate thyroid nodules; myo-inositol; selenium
MeSH Terms: conditions — Thyroid Nodule | interventions — Inositol; Selenium

STUDY DESIGN:
Intervention Model Description: One group will receive myo-inositol and selenium and one group will not be treated
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Myo-inositol and selenium supplementation (Experimental): Supplement with Myo-Inositol 600 mg + Selenium 83 mcg once a day for 6 months
  Interventions: Dietary Supplement: Myo-Inositol 600 mg + Selenium 83 mcg
- Control (No Intervention): No intervention

INTERVENTIONS:
Dietary Supplement: Myo-Inositol 600 mg + Selenium 83 mcg — Myo-Inositol 600 mg + Selenium 83 mcg: 1 tablet once a day for 6 months
  Other Names: Tiroxil 4.0
  Arms: Myo-inositol and selenium supplementation

SUMMARY:
Thyroid nodules present a variable risk of malignancy depending on the cytological result obtained from the ultrasound-assisted thyroid fine needle aspiration biopsy. According to the Italian Cytology classification SIAPEC-IAP 2014, the TIR3A nodules are indeterminate nodules with a risk of malignancy lower than 10%. Clinical and instrumental follow-up is recommended in these cases, including repetition of the fine needle aspiration.

A study have demonstrate the effect of a six-month treatment with a supplement containing myo-inositol and selenium on the size and elasticity of benign thyroid nodules.

Our hypothesis is that the use of this supplement can determine a reduction in the size and consistency of the nodule assessed through ultrasound and elastosonography also in cytologically indeterminate (TIR3A) nodules and that treatment can reduce the cellular proliferation of these nodules assessed by immunocytochemistry.

Therefore, we design a prospective randomized pilot study to assess efficacy and safety of myo-inositol and selenium in TIR3a thyroid nosules, comparing treated and untreated patients.

DETAILED DESCRIPTION:
Cytological classification of thyroid nodules (TIR 1-5) provides a useful tool in clinical practice. Each TIR class is statistically associated with a certain risk for malignancy, defining the recommended clinical action to undertake. The undetermined diagnosis (TIR 3) should represent less than 20% of patients, with an approximate risk of malignancy of 5-30%. Because of the variable risk of malignancy in the entire TIR 3 category, this is further divided into two groups: TIR 3A (low-risk follicular lesion): a heterogeneous group, with a low expected risk of malignancy (below 10%) and TIR 3B (follicular proliferation or suspected follicular neoplasia) with a higher expected risk of malignancy (15-30%). TIR3A nodules required close clinical and ultrasound follow-up and repetition of fine needle aspiration biopsy is recommended.

Selenium (Se) has the highest concentration in thyroid gland and selenium proteins are involved in thyroid hormone synthesis. Myo-inositol (MI) acts as second messengers both in thyroid differentiation and hormone synthesis and in inhibiting thyroid cells growth by inhibiting PI3K/AKT/mTOR pathway. Inositol is able to reduce NF-KB, a mediator of PI3K/AKT pathway, involved in cellular proliferation. In addition, in vitro studies demonstrated that inositol can reduce apoptosis and angiogenesis, but also inhibit the process of tumor metastasis and invasion by acting on the cytoskeleton. For this reason, this association could have a role in blocking thyroid nodule growth. Evidence from the literature highlights an important role of MI and Se in thyroid physiology and the maintenance of a euthyroid status. Particularly these micronutrients seem fundamental to counteract the onset and the worsening of thyroid alteration that could evolve into different pathological conditions if untreated. In this scenario, MI supplementation seemed to be involved also in the management of thyroidal benign nodules, with a possible effect on the size reduction. Interestingly, the administration of MI plus Se for 6 months of treatment period, was able to induce a morphological change by reducing the size and the stiffness of the nodules classified as class I or II (according to AACE/ACE/AME guidelines) in patients affected by subclinical hypothyroid.

Previous studies demonstrated a beneficial effect on subclinical hypothyroidism, restoring a euthyroid state and reducing both thyroid antibodies and TSH levels, mainly in patients affected by Hashimoto's thyroiditis. Based on these studies, nowadays, in clinical practice, oral supplementation with myoinositol and selenium is widespread and indicated in patients affected by subclinical hypotiroidism with values of TSH in the range 5-10 mcu/I with or without positivity to antibodies TPO-Ab/TG-Ab or in patients affected by Hashimoto's thyroiditis with TSH at the upper limit of the reference range.

The proposed study aims to evaluate the effect of selenium and myoinositol on possible risk factors for malignancy, as proliferation index, elastosonography characteristics (elasticity score) and TSH levels comparing a group of patients with selenium and myoinositol supplementation with a group without supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years old),
* both sexes,
* patients presenting thyroid nodules classified as TIR 3A, based on cytological evaluation on sample from the first fine needle aspiration (FNA),
* written Informed consent,
* Patients with appropriate material for subsequent immunocytochemical analysis of Ki-67 and PCNA

Exclusion Criteria:

* Patients with diagnosed thyroid malignancies of cytological diagnosis other than TIR3A
* pathological levels of the thyroid stimulating hormone (TSH) which required L-Thyroxine treatment starting
* pregnancy and/or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of differences in elastosonography after six months in patients treated with selenium and myo-inositol and patients not treated (controls) | 6 months
  Changes in elastosonographic score after treatment (comparing treated and untreated patients)- Score varies from 1 (soft) to 4 (hard)

SECONDARY OUTCOMES:
Evaluation of the inibition of the growth of thyroid nodules with Myo-inositol and Selenium supplementation | 6 months
  Changes in immunocytochemistry proliferation index (such as Ki-67 labeling index, from 0% to 100%) (comparing treated and untreated patients)
Evaluation of the differences in thyroid nodules volume in patients treated with selenium and myo-inositol | 6 months
  Changes in thyroid nodules volume (ml) in patients treated with selenium and myo-inositol (comparing treated and untreated patients)
Evaluation of the differences in thyroid hormones in patients treated with selenium and myo-inositol | 6 months
  Changes in thyroid hormones levels (TSH, FT3, FT4) in patients treated with selenium and myo-inositol (comparing treated and untreated patients)
Evaluation of the differences in anti-thyroid antibodies, in patients treated with selenium and myo-inositol | 6 months
  Changes in anti-thyroid antibodies (AbTg, AbTPO) in patients treated with selenium and myo-inositol (comparing treated and untreated patients)
Evaluation of the differences in thyroglobulin in patients treated with selenium and myo-inositol | 6 months
  Changes in thyroglobulin serum levels in patients treated with selenium and myo-inositol (comparing treated and untreated patients)
Correlation of cytological findings to histological parameters (subgroup of patients who will undergo surgical intervention) | 6 months
  Correlation of cytological findings to histological parameters

CONTACTS AND LOCATIONS:
Overall Officials: Marialuisa Appetecchia, MD, Principal Investigator — Regina Elena National Cancer Institute - IRCCS IFO
Locations (1):
- Regina Elena National Cancer Institute, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, anonymized patient data will be shared on garrbox.it repository
Supporting Information: CSR
Time Frame: After study result publication
Access Criteria: GARRbox user and working group
URL: https://gbox.garr.it/it